CLINICAL TRIAL: NCT01537471
Title: A Pilot Study of the Effects of Meclizine on Pre-Pulse Inhibition
Brief Title: The Effects of Antihistamines on Pre-Pulse Inhibition
Acronym: PPI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Wallace H. Coulter Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00028299
Record Dates: First submitted 2012-02-01; First posted 2012-02-23 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: PPI; Meclizine; Startle; Sensory processing; antihistamines
MeSH Terms: interventions — Sugars; Meclizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Other): A counterbalanced design will be used with each male subject receiving placebo and each of the anti-histamine low (12.5 mg) and high (25 mg) doses in a counterbalanced order to keep order of administration from being confounded with dose level. On one of three visits, a subject will receive placebo. The subject, study coordinator, co-investigator and outcomes assessor will remain blinded to what they received until data analysis is completed.
  Interventions: Drug: Placebo
- Meclizine (Experimental): A counterbalanced design will be used with each male subject receiving placebo and each of the anti-histamine low (12.5 mg) and high (25 mg) doses in a counterbalanced order to keep order of administration from being confounded with dose level. By the time they finish, they will have all received placebo, 12.5mg meclizine and 25mg meclizine. The subject, study coordinator, co-investigator and outcomes assessor will remain blinded to what they received until data analysis is completed.
  Interventions: Drug: Meclizine

INTERVENTIONS:
Drug: Placebo — Placebo
  Other Names: Sugar Pill
  Arms: Placebo
Drug: Meclizine — Meclizine 12.5 mg
  Other Names: Antivert, Dramamine II, Bonine, Medivert
  Arms: Meclizine
Drug: Meclizine — Meclizine 25 mg
  Other Names: Antivert, Dramamine II, Bonine, Medivert
  Arms: Meclizine

SUMMARY:
The purpose of the investigators research is to test whether problems people have with processing their senses (feeling overwhelmed, distracted or upset by sounds and other stimuli) can be lessened by meclizine, a drug found in many over the counter antihistamines, which are medicines used for things like allergies, sleep problems, or the common cold.

DETAILED DESCRIPTION:
This experiment will test the efficacy of acute anti-histamine doses on the acoustic startle response and prepulse inhibition (or PPI, a well-known neurobehavioral phenomenon used to characterize sensorimotor modulation described in detail below) in a male population with high baseline sensory startle levels. In addition, sex differences in baseline PPI (i.e. without anti-histamine administration) in subjects of this population will be investigated.

The main hypothesis of the study is that the H1¬-antagonist meclizine will be effective in restoring low levels of PPI observed in the subject pool so that sensory gating is made more effective. The dependent measures will be startle response magnitude and pre-pulse inhibition.

The experiment will take place in four sessions, carried out on different days. Consecutive test sessions will take place no earlier than 3 days, and no longer than 21 days apart. Before being recruited into the study, potential participants will go through a phone screen-a pre-experiment screening questionnaire (separate) to exclude subjects with neurological disorders, certain psychiatric disorders, who smoke or use nicotine products, or who use certain drugs (see exclusion criteria below) as they can affect PPI levels. If they are eligible per the phone screen, subjects will come in for screening (test day 1). They will be again asked about their tobacco/nicotine use and what medications they are currently taking. They will be asked about their caffeine history use. Caffeine and caffeine withdrawal both have effects on startle response but not on PPI so we are not restricting subject's caffeine use, but collecting this information. CO levels will be collected using a CO monitor to confirm that participants have not recently used a tobacco product. They will be asked questions about psychiatric symptoms, personality, and how they cope with stress. Participants' startle responses and PPI will be tested in the laboratory (see below).

During the following three test days (2-4) before dispensing study drug, male participants who qualify, will be asked to fill out a questionnaire about tobacco or nicotine use since their previous visit along with assessing any change in their medications (specifically verifying that a male participant has not used an allergy, cold/flu medication within 3 days of their study visit). If the participant answers yes to either question, they will be asked to return to the clinic on a different day: 1) 3 or more days post using an antihistamine or 2) at least 2 weeks post using tobacco or nicotine. Both antihistamine medications or tobacco/nicotine recent use can effect a participant's PPI which is why we have the need to ask male participants about any possible changes. They will also be asked how they arrived to the clinic to verify that they have a driver who came with them/dropped them off, had a hired driver provided by the study if they live in Durham or came by bus or by foot. They will be asked about their caffeine use on the day of their experiment. Their baseline sedation level will be assessed. On test days 2-4, the test procedure employed on test day 1 will be repeated, but 60 minutes before the start of each test sessions, participants will receive a placebo, a low (12.5 mg) dose of meclizine, or a high (25 mg) dose of this drug in a counterbalanced order.

Male participants (n = 20) will receive the study medication or placebo orally and will be provided water at administration at visits Day 2-4. Placebo and meclizine capsules will be identical in shape, size, and color. The randomization and counterbalancing of the order of dosing will be in charge of Dr. Levin. In order to ensure that the blind procedure is not violated, Dr. Levin (a) will provide the identical capsules for the study to the Study Coordinator in containers labeled "Subject X, day Y", and (b) will have no contact with the participants in the study. Meclizine and placebo will be dispensed by the Study Coordinator under the administrative supervision of Dr. Rosenthal, and under the clinical supervision of a study physician. During the resting period between pill ingestion and the experimental task, male participants will be asked to sit in a lab room and read or use the internet. At 20 minutes and 40 minutes post drug, sedation level will be assessed using the scale listed below.

In each PPI test session throughout all 4 visits, male participants will begin with a resting baseline period of 5 minutes, where they will be asked to sit quietly and still in a sound and temperature controlled lab room, with their eyes open looking at a fixation cross on the monitor. Baseline is conducted to obtain measures of emotional arousal and sedation prior to the experimental manipulations. As such, during baseline psychophysiological measures will be collected. Self-reported emotional arousal will be obtained at the beginning and end of the baseline period using the Self-Assessment Manikin (Bradley, 1999), which assesses arousal and valence of affective state using Likert (1-9) scales. Self-reported level of sedation will be assessed at the same time points as emotional arousal (using a modified Self-Assessment Manikin using the same Likert 1-9 scale). Next, participants will be exposed to an initial adaptation phase, in order for them to become acquainted with the startle stimuli (pulses and prepulses), and their startle responses reach a stable level. In this phase, 4 blocks of prepulse-pulse (pP) and pulse-alone (P) trials will be presented, with an inter-trial interval (ITI) of 20 seconds (+/- 5 sec). After the initial adaptation phase, participants will be instructed to view a computer monitor where random geometric figures will be presented, while simultaneously 10 blocks of auditory pP and P trials will be presented with an ITI of 20 sec. Each test session will last around 15 minutes. At the end of the test session, the standardized lab test to assess the participants' attention level described above will be presented again.

Females will only complete the first day of testing (in the same way as described for male subjects above).

ELIGIBILITY:
Inclusion Criteria:

* 18-40 males or females
* Startle response >0.5
* PPI < 32
* CO level <8ppm

Exclusion Criteria:

* Tobacco or nicotine use within 2 weeks of screening
* Current or history of a neurological disorder of neurological event
* Negative response to antihistamine use in past
* ECT treatment in the past 6 months
* Current or past history of manic or hypomanic episodes (SCID-I)
* Current or history of psychotic disorder
* Current alcohol or substance abuse/dependence
* Positive urine drug test
* CO level of >8ppm
* Startle <0.5 & overall PPI >32 (assessed during study)
* Significant hearing problem

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in PPI | Screening Day 1, Days 2-4
  The primary outcome will measure change in subjects' PPI depending on whether they were given meclizine during the study. Prepulse inhibition (PPI) of the startle reflex by a weak pre-pulse will be assessed during each laboratory session. It is measured using electromyographic (EMG; i.e., for assessing eye blink magnitude) responses.

SECONDARY OUTCOMES:
Sedation | Day 2, Day 3, & Day 4
  A Baseline sedation level at the beginning of each visit will be collected. Then study drug (meclizine/placebo) will be given and a sedation level will be collected at 20 minutes and 40 minutes post drug as well as during the PPI experiment pre & post. The Sedation scale will be used (a modified version of the SAM scale).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Z Rosenthal, PhD, Principal Investigator — Duke University; Ed Levin, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Braff D, Stone C, Callaway E, Geyer M, Glick I, Bali L. Prestimulus effects on human startle reflex in normals and schizophrenics. Psychophysiology. 1978 Jul;15(4):339-43. doi: 10.1111/j.1469-8986.1978.tb01390.x. No abstract available. PMID 693742
- [Background] Castellanos FX, Fine EJ, Kaysen D, Marsh WL, Rapoport JL, Hallett M. Sensorimotor gating in boys with Tourette's syndrome and ADHD: preliminary results. Biol Psychiatry. 1996 Jan 1;39(1):33-41. doi: 10.1016/0006-3223(95)00101-8. PMID 8719124